CLINICAL TRIAL: NCT01479166
Title: Bronchial Inflammation of Small Airways in Patients With Cystic Fibrosis
Acronym: FRA-MUKO
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Stefan Zielen, Professor Dr. med. Stefan Zielen, Johann Wolfgang Goethe University Hospital
Other Study IDs: 85/11
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; HRCT; Sputum; Blood; Inflammation; adaptive immune system; innate immune system
MeSH Terms: conditions — Cystic Fibrosis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum and Sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- affected patients with small airway disease (SAD): 20 patients suffering from mild cystic fibrosis and involvement of small airways
- affected patients without small airway disease (SAD): 20 patients suffering from mild cystic fibrosis without SAD
- non-affected patients: 20 matched controls not suffering from cystic fibrosis

SUMMARY:
In the planned study, 60 patients with mild cystic fibrosis (CF) with and without the involvement of small airways (small airway disease - SAD) are to be compared with a historical control group matched in age and gender. During the first study visit subjects are asked to perform a pulmonary function test (spirometry, body plethysmography with helium, determination of "Trapped Air") and exhaled nitric oxide (eNO) and exhaled carbon monoxide (eCO) measurements will be done in exhaled air. In addition, a blood sample is drawn to describe inflammatory status. Sputum is induced as well. During the second study visit, a non-specific bronchial provocation test(methacholine PD20 FEV1) is performed.

The aim of the study is to get a characterization of the bronchial and systemic inflammation (IL-1ß, IL-6, IL-8, IL-17, TNF-α, NFKB, and recognition structures like TLR2 and TLR4) in CF patients with and without the involvement of the small airways, which may point to new treatment strategies.

DETAILED DESCRIPTION:
Aim of this study is the characterization of patients with mild cystic fibrosis in terms of lung function, bronchial hyperreactivity and the degree of systemic and bronchial inflammation.

Sputum and serum samples are analyzed by quantitative real-time polymerase chain reaction(qRT-PCR) and by cytometric bead assay (CBA). Components of the innate immune system (mannose-binding protein, TLR recognition proteins and surfactant proteins) are genetically determined from sputum or blood respectively. In order to support the analyzed lung function and sputum/ serum biomarker data the investigators will also rely on pre-existing imaging data like chest x-rays or high-resolution computer tomography (HRCT)of the lungs.

Methods and Work Programme:

This study consists of two study visits (V1 and V2)

V1:

Measurement of nitric oxide in exhaled air (eNO) Measurement of carbon monoxide in exhaled air (eCO) Lung function testing with spirometry and body plethysmography Blood test: blood count, CRP, RAST, serum inflammatory mediators, genetic markers of the non-specific pulmonary defense system Induced sputum for inflammatory mediators and microbiological investigations

V2:

Unspecific bronchial provocation test with methacholine (PD20 FEV1 methacholine) Lung function testing with spirometry and body plethysmography

Study population:

CF Children and adults (6 - 60 years of age) and a healthy control group (6-60 years of age). Both patients and healthy subjects are recruited from the Christiane Herzog Cystic fibrosis outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* confirmed diagnosis of CF (known mutations and/or sweat chloride test > 60mval/l)
* age between 6 and 60 years
* vital capacity > 75%
* Ability to perform lung function tests and inhalation

Exclusion Criteria:

* < 6 and > 60 years of age on the day of written informed consent
* Acute illness with systemic or bronchial inflammation
* every chronic condition or infection (eg HIV, tuberculosis, malignancy)
* pregnancy
* known alcohol and/ or drug abuse
* Inability to understand the extent and scope of the study
* Participation in another study

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study is carried out in CF children and adults (6 to 60 years) and healthy controls (6-60 years). Both patients (40) and healthy subjects (20) are recruited from the Christiane Herzog CF outpatient clinic of Johann Wolfgang Goethe-University, Frankfurt/M, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Bronchial Inflammation in sputum of patients with CF | 24 months
  Measuring IL-8 in induced sputum compared to induced sputum of age matched controls

SECONDARY OUTCOMES:
Inflammatory proteins like (Il-1,IL-6, TNF alpha) in induced sputum | 24 months
  Measuring secondary parameters in induced sputum by cytometric bead assay

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zielen, MD, PhD, Principal Investigator — Children´s Hospital of Johann Wolfgang Goethe-Univeristy, Frankfurt/Main
Locations (1):
- Children's Hospital, Johann Wolfgang Goethe-University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Background] Eickmeier O, Huebner M, Herrmann E, Zissler U, Rosewich M, Baer PC, Buhl R, Schmitt-Grohe S, Zielen S, Schubert R. Sputum biomarker profiles in cystic fibrosis (CF) and chronic obstructive pulmonary disease (COPD) and association between pulmonary function. Cytokine. 2010 May;50(2):152-7. doi: 10.1016/j.cyto.2010.02.004. Epub 2010 Feb 23. PMID 20181491
- [Background] Tiddens HA, Donaldson SH, Rosenfeld M, Pare PD. Cystic fibrosis lung disease starts in the small airways: can we treat it more effectively? Pediatr Pulmonol. 2010 Feb;45(2):107-17. doi: 10.1002/ppul.21154. PMID 20082341